CLINICAL TRIAL: NCT06149793
Title: Empagliflozin in CFRD: Efficacy and Safety of SGLT2 Inhibitor Therapy in Overweight and Obese Subjects With Cystic Fibrosis-related Diabetes: a Pilot Study
Brief Title: SGLT2 Inhibitor Therapy in Cystic Fibrosis-related Diabetes
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MED-2023-31645
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis-related Diabetes; Cystic Fibrosis
Keywords: CFRD; cystic fibrosis; cystic fibrosis related diabetes; empagliflozin
MeSH Terms: conditions — Cystic Fibrosis | interventions — empagliflozin; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Intervention Model Description: This will be a placebo-controlled, randomized, double blind, crossover study with a 4 week wash out period.
  Collect pilot data on the safety, tolerability, and feasibility of empagliflozin therapy in overweight/obese patients with CFRD to support a future larger randomized controlled trial.
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- empagliflozin (Active Comparator): randomized to study medication (empagliflozin) 10 mg taken by mouth daily for 4 weeks
  Interventions: Drug: Empagliflozin
- placebo control (Placebo Comparator): randomized to placebo control taken by mouth daily for 4 weeks
  Interventions: Other: Placebo Control

INTERVENTIONS:
Drug: Empagliflozin — Sodium glucose co-transporter 2 inhibitor
  Other Names: Jardiance; SGLT2 inhibitor
  Arms: empagliflozin
Other: Placebo Control — Placebo Control
  Arms: placebo control

SUMMARY:
This will be a placebo-controlled, randomized, double blind, crossover study with a 4 week wash out period.

Collect pilot data on the safety, tolerability, and feasibility of empagliflozin therapy in overweight/obese patients with CFRD to support a future larger randomized controlled trial.

DETAILED DESCRIPTION:
The overall goal of this proposal is to collect pilot data for safety and feasibility metrics to support a future larger randomized controlled trial. In this study, we will examine the safety and tolerability of Sodium glucose co-transporter 2 inhibitor (SGLT2i) empagliflozin as an add-on therapy to insulin for overweight/obese adult patients with CFRD. We hypothesize that empagliflozin will be safe, well tolerated and will improve glycemic control in overweight/obese adult patients with CFRD.

Specific Aim 1: Collect pilot data on the safety, tolerability, and feasibility of empagliflozin therapy in overweight/obese patients with CFRD to support a future larger randomized controlled trial.

Hypothesis 1: Empagliflozin will be safe and well tolerated, with no evidence for electrolyte abnormalities, metabolic acidosis, ketosis or increased risk of severe hypoglycemia in overweight/obese adults people with CFRD.

Specific Aim 2: Collect preliminary data to evaluate the effect of empagliflozin on glycemic outcomes.

Hypothesis 2: Treatment with empagliflozin will improve glycemic control as indicated by glucose levels as measured by oral glucose tolerance test (OGTT), and on glycemic outcomes as measured by continuous glucose monitoring (CGM).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 18 years or older with CFRD and on insulin treatment
* BMI >25 kg/m2
* A participant who is capable of becoming pregnant must agree to take precautions that are effective in preventing pregnancy throughout this study. These methods could include one of the following 1. Complete abstinence from sexual intercourse; 2. Tubal ligation; 3. Use combination of two forms of contraception during the study including, oral, injectable, or implanted hormonal contraceptives, intrauterine device or barrier method.

Exclusion Criteria:

* acute pulmonary exacerbation requiring IV antibiotics or systemic glucocorticoids within 4 weeks prior to baseline study procedures
* less than 12 weeks since start of a new CFTR corrector/modulator therapy
* type 1 diabetes
* Positive GAD 65 antibody or low fasting C-peptide (below the normal reference range of the lab)
* A history of diabetic ketoacidosis
* history of recurrent genital or urinary tract infections
* pregnancy or lactation
* prior solid organ transplant
* Chronic liver disease (based on problem list in medical records or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times elevated above the upper limit of normal.
* chronic kidney disease (eGFR < 60mL/min/1.73 m2)
* Hypersensitivity to empagliflozin or any excipients of Jardiance
* History of eating disorder
* Non-English speakers and those unable to read in English • Diminished capacity to consent (study staff will utilize the MacCAT-CR for assessment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility, safety, tolerability | Duration of anticipated participation for an individual participant's would be around 15 weeks.Duration anticipated to complete all study procedures, including any long-term follow-up, and data analysis is 24 months.
  The primary outcomes are related to feasibility, including safety and treatment tolerability. Safety will be evaluated as the proportion (in %) of participants who experience a serious adverse event during the study. Tolerability will be evaluated as the proportion (in %) of participants who discontinue their assigned treatment due to side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No